CLINICAL TRIAL: NCT01551797
Title: A Proof of Principal Study to Investigate the Pharmacokinetic Profiles of Sustained Release and Standard Paracetamol Formulations
Brief Title: A Pharmacokinetic Study to Compare Sustained Release and Standard Paracetamol Formulations.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A2750894
Record Dates: First submitted 2012-02-23; First posted 2012-03-13 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Test Sustained Release (SR) Paracetamol (2000 mg) (Experimental): A single 2000 mg oral dose of SR paracetamol formulation (2 x 1000 mg) administered with 150 mL of water.
  Interventions: Drug: Paracetamol 1000 mg
- Test SR Paracetamol (1500 mg) (Experimental): A single 1500 mg oral dose of SR paracetamol formulation (2 x 750 mg) administered with 150 mL of water.
  Interventions: Drug: Paracetamol 750 mg
- Reference Paracetamol (2000 mg) (Active Comparator): Two single 1000 mg doses of paracetamol (2 x 500 mg/dose) administered orally 6 hours apart, administered with 150 mL of water.
  Interventions: Drug: Paracetamol 500 mg

INTERVENTIONS:
Drug: Paracetamol 500 mg — Standard Paracetamol formulation
  Arms: Reference Paracetamol (2000 mg)
Drug: Paracetamol 1000 mg — Paracetamol Sustained Release formulation
  Arms: Test Sustained Release (SR) Paracetamol (2000 mg)
Drug: Paracetamol 750 mg — Paracetamol Sustained Release formulation
  Arms: Test SR Paracetamol (1500 mg)

SUMMARY:
This proof of principle study will evaluate an experimental formulation of paracetamol that is being developed for eventual long lasting use. This study is also used for drug safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI): Body Mass Index must be in the range 19-28 kg/m2.

Exclusion Criteria:

* Disease: Current or recurrent disease that could affect the action, absorption, elimination or disposition of the study medication or clinical or laboratory assessments (e.g. hepatic disorders evidenced by abnormal liver function test, hepatitis serology test and liver image studies, renal insufficiency, congestive heart failure).
* Current or relevant previous history of serious, severe or unstable physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the study medication or procedures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Median time to reach therapeutic plasma concentration of paracetamol | Baseline, 15 min, 30 min, 45 min, 1, 1.5 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 14, 15, 16, and 18 hours post-treatment
  Time period in hours over which plasma paracetamol concentration is elevated at or above 4 micrograms (μg)/milliliter (mL).

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve (AUC) | Baseline, 15 min, 30 min, 45 min, 1, 1.5 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 14, 15, 16, and 18 hours post-treatment
  Area under the plasma concentration-time curve from zero to 6 hours (AUC 0-6 hours), 12 hours (AUC 0-12 hours) to be determined. AUC0-t : the area under the plasma concentration-time curve from zero to time t when paracetamol remains detectable. AUC0-∞: the area under the plasma concentration time curve from zero and extrapolated to infinity time.
Time to maximum plasma concentration (Tmax) | Baseline, 15 min, 30 min, 45 min, 1, 1.5 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 14, 15, 16, and 18 hours post-treatment
  Tmax for paracetamol to be determined.
Half-life of elimination (T 1/2) | Baseline, 15 min, 30 min, 45 min, 1, 1.5 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 14, 15, 16, and 18 hours post-treatment
  T 1/2 of paracetamol to be determined.
Elimination rate (Kel) | Baseline, 15 min, 30 min, 45 min, 1, 1.5 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 14, 15, 16, and 18 hours post-treatment
  Kel of paracetamol to be determined.
Maximum plasma concentration (Cmax) | Baseline, 15 min, 30 min, 45 min, 1, 1.5 2, 3, 3.5, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 10.5, 11, 11.5, 12, 12.5, 13, 14, 15, 16, and 18 hours post-treatment
  Cmax of paracetamol to be determined.
Number of participants with Adverse Events (AEs) and Serious AEs | Day 1 through Day 14 (follow-up visit)
  Safety evaluation

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Charles River Clinical Services Northwest, Inc., Tacoma, Washington, United States